CLINICAL TRIAL: NCT06110338
Title: A Phase 1, Double-blind Study to Evaluate the Safety and Tolerability of a Single-dose Administration of IBI355 in Health Adults
Brief Title: Safety and Tolerance Study of IBI355 in Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI355A101CN
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- IBI355 dose 1 (Experimental): IBI355 0.3mg/kg and placebo will be given to the subjects (3:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose 4 (Experimental): IBI355 7.5mg/kg and placebo will be given to the subjects (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose 6 (Experimental): IBI355 25mg/kg and placebo will be given to the subjects (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose 7 (Experimental): IBI355 35mg/kg and placebo will be given to the subjects (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose 2 (Experimental): IBI355 1mg/kg and placebo will be given to the subjects (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose 3 (Experimental): IBI355 3mg/kg and placebo will be given to the subjects (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose 5 (Experimental): IBI355 15mg/kg and placebo will be given to the subjects (6:2)
  Interventions: Drug: placebo; Drug: IBI355

INTERVENTIONS:
Drug: placebo — placebo iv. once.
Drug: IBI355 — IBI355 iv. once.

SUMMARY:
This study is being done to find out if IBI355 is safe and tolerance in health volunteers. The study will test increasing single doses of IBI355 given to adult health volunteers. The goal is to confirmed the safety of the highest dose of IBI355 or to find out the highest dose of IBI35 that can be given to health volunteer that dose not cause unacceptable side effects. Different dose regimens will be evaluated. The pharmacokinetics and ADA of IBI355 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have decided to voluntarily participate in the study and provided a written consent regarding observance of precautions after having been informed of and having fully understood the objectives, methods, and effects of the study in detail;
2. Healthy male and female aged 18 years or above ;
3. Subject with a Body Mass Index (BMI)* between 18.5 and 28.0 kg/㎡;
4. subjects with a normal laboratory examination，ECG， X-ray.

Exclusion Criteria:

1. Subjects with a history of allergy；
2. Subjects participated in the other clinical trail in 1 month or less than 5 t1/2 since the previous clinical trial (which is longer)；
3. Subjects with an infection requiring systemic medication was present within 30 days prior to randomization;
4. HIV-Ab、RPR、HCV-Ab、HBV、HBeAg or HBcAb, one of them positive;
5. There have a clinical or imaging evidence that the subject with active tuberculosis, or there is evidence that the subject is in the incubation period for tuberculosis;
6. Patients with a history of central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders and other systemic diseases;
7. Subject with a hcg positive;
8. Patients with a history of neuropsychiatry or who are considered unfit to participate in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Incidence of AE、SAE after receiving IBI 355 | week 0-12

SECONDARY OUTCOMES:
Area Under Curve, (AUC）、Maximum serum concentration of drug(Cmax）、Clearance (CL）、Apparent volume of distribution(V） and Half- life(t1/2）of IBI355 | week 0-12

CONTACTS AND LOCATIONS:
Locations (1):
- Aerospace Center Hospital, Beijing, Beijing Municipality, China